CLINICAL TRIAL: NCT00575003
Title: Double-Blind, Placebo-Controlled Study to Investigate an Immunomodulatory Therapy (CYT003-QbG10) in Adult Patients With Perennial Allergic Rhinoconjunctivitis
Brief Title: Study to Investigate an Immunomodulatory Therapy in Adult Patients With Perennial Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytos Biotechnology AG (Industry)
Responsible Party: Dr. Philipp Mueller, Cytos Biotechnology AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYT003-QbG10 08
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Perennial Allergy to House Dust Mite and/or Cat
MeSH Terms: interventions — CYT003-QbG10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CYT003-QbG10
- 2 (Placebo Comparator)
  Interventions: Drug: CYT003-QbG10

INTERVENTIONS:
Drug: CYT003-QbG10 — 6 subcutaneous injections

SUMMARY:
The purpose of the study is to test the efficacy of a vaccine against house dust mite and/or cat allergy compared to placebo in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate perennial allergic rhinoconjunctivitis due to hypersensitization towards house dust mite and/or cat allergens

Exclusion Criteria:

* Clinical relevant other allergies (perennial or seasonal) that could potentially interfere with the patient's study treatment schedule or assessments.
* Use of any concomitant medication that could affect the patient's study treatment response or assessment results.
* Any clinically relevant concomitant disease as judged by the investigator.
* Pregnancy or female planning to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Conjunctival provocation test with allergen and rhinoconjunctivitis symptoms in daily life | on 4 occations over 1 year

SECONDARY OUTCOMES:
Safety and tolerability of the vaccine by collection of adverse events | at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Audra Blaziene, Principal Investigator — Vilnius University Hospital
Locations (7):
- Estonia (2):
  - Tartu University Clinic, Out-Patients Department, Tartu
  - Tartu University Clinic, Lungs Clinic, Tartu
- Latvia (2):
  - The centre of the investigation in treatment of allergic disease, Riga
  - SNC Uniclinica, Riga
- Lithuania (3):
  - Kaunas County Hospital, Department of Pulmonology and Allergology, Kaunas
  - Kaunas Medical University Hospital, Department of Pulmonology and Immunology, Kaunas
  - Vilnius University Hospital, Centre of Pulmonology and Allergology, Vilnius